CLINICAL TRIAL: NCT00427180
Title: Extended Pilot Study to Evaluate Pattern Recognition With a Chronic Retinal Implant System
Brief Title: IRIS PILOT - Extended Pilot Study With a Retinal Implant System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Intelligent Medical Implants GmbH (Industry)
Responsible Party: Intelligent Medical Implants GmbH, Medical device industry
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-80-00-00-00-01-V01; SP-80-00-00-00-02-V01 (Other: IMI Intelligent Medical Implants GmbH); SP-80-00-00-00-03-V01 (Other: IMI Intelligent Medical Implants GmbH)
Record Dates: First submitted 2007-01-25; First posted 2007-01-26 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Retinitis Pigmentosa; Cone-Rod Dystrophy; Choroideremia
Keywords: Visual Perception; Retina; Light; Retinitis Pigmentosa; Visual acuity; Retinal Implant; Electrical stimulation
MeSH Terms: conditions — Retinitis Pigmentosa; Cone-Rod Dystrophies; Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Retinal Implant System (IRIS) — AIMD - Active Implantable Medical Device designed for artificial electrical neural stimulation of photoreceptor degenerated retina
  Other Names: IRIS

SUMMARY:
Investigate whether blind subjects that fulfil the patient criteria provided with a Retinal Implant are able to differentiate between simple patterns like horizontal bar, vertical bar and cross.

DETAILED DESCRIPTION:
The Retinal Implant System consists of three main components, the Retinal Stimulator, which is the component actually implanted into the eye, the visual interface, and the Pocket Processor The Retinal Stimulator will be implanted into the eye of a blind subject during a surgical operation. However, the external components are activated only during the test sessions under the control of the investigator team. In a first step of the investigation a software controlled system on a PC which is connected to the Pocket Processor via Ethernet interface, will generate the defined stimulation patterns (bars, crosses, cubes). During the test session, the blind subject is exposed to a series of these stimulation patterns and he / she has to describe the visual perceptions. Based on his descriptions and in an interactive way, the stimulation signal is subsequently be modulated by changing parameters like amplitude, duration of impulse, polarity, number of repetitions or pulse frequency on the PC.

In a second step the visual interface is equipped with a camera which presents realtime images to the subject. Data obtained from the investigation with computer generated patterns in the first step are used in the second step to improve the fitting software for the use in the camera supported system.

Finally the system should enable the subject to recognize simple images supported from the camera.

ELIGIBILITY:
Inclusion Criteria

* Age between 30 and 79 years at the date of enrollment
* Normal hearing and linguistic understanding (with hearing aids if - necessary and in the language of the hospital or in English)
* Ability to understand the study and procedures involved
* Willingness to participate and comply with follow-up procedures
* Good general health based on investigator's opinion
* Ability to undergo surgery using general anaesthesia
* Signed informed consent
* RP, choroideremia, or rod cone dystrophy
* Visual field less than 40 ° (if measurable)
* Visual acuity not better than (1/50), (logMAR≥1.7)
* Visual function stable for a duration of at least one year (according to subject statement)
* Normal eye pressure (9-21 mmHg)
* Bulbus length (AP) between 21 and 25 mm

Exclusion Criteria

* Allergic response to multiple antibiotics
* Known allergies to materials of the implant
* Known carrier of multi-resistant organisms
* Pregnancy or lactating
* History of epileptic seizures
* Having active implantable devices (or need within the next 3 years)
* Patients with cancer or patients received cancer therapy within the last 2 years
* Currently undergoing psychiatric treatment without expert opinion approving participation on the study
* Patients having insufficient mental capacity
* Neurological diseases, in particular those affecting nerve conduction velocities
* Patients currently taking medications affecting brain function
* Immunosuppressive subjects

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Investigate whether blind subjects that fulfill the patient criteria provided with a Retinal Implant are able to differentiate between simple patterns like horizontal bar, vertical bar and cross. | 18 months

SECONDARY OUTCOMES:
Secondary goals of this study phase are: Further evaluation of stimulation parameters, Light localization with use of camera, Safety verification of stimulation parameters | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gisbert Richard, Prof., Principal Investigator — Klinik und Poliklinik für Augenheilkunde Hamburg-Eppendorf

REFERENCES:
- [Background] Hornig R, Laube T, Walter P, Velikay-Parel M, Bornfeld N, Feucht M, Akguel H, Rossler G, Alteheld N, Lutke Notarp D, Wyatt J, Richard G. A method and technical equipment for an acute human trial to evaluate retinal implant technology. J Neural Eng. 2005 Mar;2(1):S129-34. doi: 10.1088/1741-2560/2/1/014. Epub 2005 Feb 22. PMID 15876648